CLINICAL TRIAL: NCT01828372
Title: Quantification of Drugs and Their Metabolites in Patients at the Cologne University Hospital
Brief Title: Quantification of Drugs and Their Degradation Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Ali Mohammad Nejad Sigaroudi, Medical Doctor, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: KPUK-12-GenPOPPK-2; 2013-000779-33 (EudraCT Number)
Record Dates: First submitted 2013-03-14; First posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Liver Insufficiency; Kidney Failure, Chronic; Obesity; Pregnancy; Breast Feeding, Exclusive; Sepsis; Multiple Organ Failure
Keywords: concomitant diseases; multiple drug consumption; therapeutic drug monitoring; TDM; drug monitoring; drug level; quantification; drug; drug concentration; concentration; therapeutic range; therapeutic index
MeSH Terms: conditions — Hepatic Insufficiency; Kidney Failure, Chronic; Obesity; Breast Feeding; Sepsis; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- additional blood withdrawals (Other): Theoretical anyone with taking a drug of interest (see "list of substances and metabolites of interest") can join this trial. But we turn mainly our attention to patient groups who are excluded in modern drug approval studies.
  Interventions: Other: additional blood withdrawals

INTERVENTIONS:
Other: additional blood withdrawals — Blood withdrawals by either venous puncture or placement of permanent venous catheter.

SUMMARY:
The study includes two study parts in which blood is collected from the patients.

Study part A (observational study, already received positive ethics committee vote; Our sign: 12-330): Use of blood samples gathered during routine blood withdrawal Study part B (interventional study in the sense of additional blood samples but without an investigational product): Optional, for further pharmacokinetic questions: blood withdrawal with a maximum of 20 ml ( ten tubes of 2 ml each) within a maximal study length of four weeks.

The primary objective of this study is to gain an overview about drug concentrations in plasma and/or cerebrospinal fluid (CSF), in order to determine pharmacokinetics of drugs in patients. Any drug may be tested, however the initial focus is on antiinfective, antineoplastic, and antipsychotic drugs.

Many published studies show that there is a profound lack of information on pharmacokinetics and interactions of many commonly used drugs in clinical routine, and that drug concentrations, if controlled by therapeutic drug monitoring, are not in the therapeutic range (provided that such ranges are known at all).

DETAILED DESCRIPTION:
For an effective pharmacotherapy in patients with different demographic characteristics (age, weight or lean body mass), there is often a lack of information on the dosage of drugs.

The predictability of the action of a drug is additionally impaired by genetic predisposition. Even if the effect of genetic variants has been demonstrated, the respective characteristic for the patient is usually not known.

For example, a study (Gamelin et al., 2008) of the "old" cytostatic drug 5-fluorouracil shows its genetically-dependent efficacy.

Only in about one third of patients does the concentration reach the desired therapeutic range (the dosage adjusted to body surface).

There is a significant lack of information on the pharmacokinetics, especially in critically ill patients.

These patients are excluded in modern drug approval studies, although it is anticipated that, depending on the drug, many patients with severely impaired renal function, renal replacement therapy, severe hepatic dysfunction, sepsis or multiple organ failure may later on obtain the substance.

This knowledge gap on the specific pharmacokinetics of drugs in selected populations is present not only for new drugs, but also for those that have already been used in therapy for decades.

Particularly for the effect of body weight and liver function on pharmacokinetics, data is very sparse. For the latter, the lack of data is particularly striking, when searching for data concerning patients with severe hepatic dysfunction. If occasional data for specific drugs are available, then for most substances these are not sufficient to develop a safe dosing regimen, e.g. for the aforementioned example of 5-fluorouracil. Furthermore, for many drugs reliable pharmacokinetic data in renal impairment or renal replacement therapy are not available. The available data is generally much better than in hepatic insufficiency, but especially the lack of data on the pharmacokinetics of metabolites in renal insufficiency may be of relevance, as such metabolites are active and play an important role for the effect, but they may also be responsible for side effects. To illustrate, the "Fachinformation" (as of April 30th 2012), the legally binding document for dosing issues of drugs in Germany, is attached. This table provides a selection of important drugs, while it is not exhaustive.

In hospitals predominantly severely ill patients are treated and several drugs are administered simultaneously. Thus, the issue of drug-drug interaction is in the center of attention. Unexpected new clinical interactions of drugs known for a long time, or interactions of well-known substances with new substances are reported. A recent example is an interaction caused by Cotrimoxazol, a drug combination used for decades (Antoniou et al., 2011).

In summary, it can be stated that in drug therapy there is a high demand for both the quantification of in vivo plasma and liquor drug concentrations and quantifying the effect of different characteristics on the pharmacokinetics of the drugs. Thus, concentrations for a broad range of substances which are used in the Cologne University Hospital should be measured, including their respective metabolites. Concentrations both in plasma and in CSF (for drugs supposed to have an effect on the central nervous system) will be quantified. This screening approach is possible due to the increasing availability of highly sensitive and selective liquid chromatography - tandem mass spectrometry (LC-MS/MS) methods, thereby the number of measurable substances markedly increased. The initial focus of our project is on the antiinfective, antineoplastic and antipsychotic agents.

ELIGIBILITY:
Inclusion Criteria:

* Both genders are included.
* Patients willing and capable to confirm written consent prior to enrolment after ample information was given are eligible for the study.

Exclusion Criteria:

* In Study Part B patients with hemoglobin less 7 mg/dl or less 10 mg/dl including serious symptoms of anemia such as increased heart rate, shortness of breath, dizziness, weakness etc.
* The hemoglobin value must not be 10 days or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-04 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Outcome Measures (e.g., Cmax, AUC) | within four weeks after administration of drug of interest
  These assessments rely on multiple measurements over time and the Time Frame may include multiple time points describing the interval at which data are collected

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Fuhr, Professor, Study Director — Department of Pharmacology
Locations (1):
- Department of Pharmacology, Cologne University Hospital, Cologne, North Rhine-Westphalia, Germany